CLINICAL TRIAL: NCT07099508
Title: Factors Influencing Home Nursing Care Service: a Pilot Study Shedding Light Over the Feasibility
Brief Title: Factors Influencing Home Nursing Care Service
Acronym: HoNuCaS-01
Status: Not yet recruiting | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: Azienda Ulss 6 Euganea (Other)
Responsible Party: Sponsor
Other Study IDs: HoNuCaS-01
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Home Care Services
Keywords: Home Nursing Care; Nursing time measurement; Travel time; Health planning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This pilot study investigates the feasibility of a prospective longitudinal observational approach to identify variables influencing home nursing care time. Conducted within the ULSS 6 Euganea health district in Italy, the study will analyze nursing care and travel time across approximately 350 home visits involving up to 200 voluntarily enrolled adult patients. Data will be collected anonymously by nurses using a digital tool (REDCap), capturing a predefined core set of variables previously selected via the Delphi method. The study aims to understand the association between individual, contextual, and organizational variables and the time required for home nursing interventions. Results will inform better planning and resource allocation for home care services.

ELIGIBILITY:
Inclusion Criteria: all patients receiving home care nursing services who agree to voluntary participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving home care nursing services:
  * Condition of frailty or dependence: often associated with chronic or degenerative diseases.
  * Presence or absence of family support network: the lack of caregivers can increase the required frequency of visits.
  * Multimorbidity: patients often suffer from multiple chronic conditions (e.g., diabetes, heart failure, COPD, dementia).
  * Disabilities or functional limitations: motor, sensory, or cognitive impairments that necessitate home-based care.
  * Ongoing or complex healthcare needs: including advanced wound care, stoma management, enteral/parenteral nutrition, intravenous therapy.
  * End-of-life or palliative care: some patients receive home palliative care (e.g., type III Integrated Home Care).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Factors thath influence home care nurses | From the enrollment to the end of the study at two months
  Measure the factors that influence the work of home care nurses in individual subjects and different territorial contexts in relation to care time.
  * patient's socioeconomic status (age, level of education, understanding of italian language, rural or urban context,..)
  * patient's clinical status (hospitalizations, type of assistance needed, type of support, diagnosis, mobility status..)
  * caregiver (type, hours of formal and informal caregiving, coping, knowledge of the patient's medical history,..)
  * visit specific variables (presence of animals, number of services provided, time required for the service in minutes,..)
  * IDC-PAL items

SECONDARY OUTCOMES:
Time and space spent by the nurse traveling to the patient's home | From the enrollment to the end at two months
  Travel times in minutes and distance traveled in Kilometers, calculated by the nurses from departure to arrival at each patients' home.

IPD SHARING:
Plan to Share IPD: Undecided